CLINICAL TRIAL: NCT00566904
Title: Phase 1 Novel Topical Treatment for Post-herpetic Neuralgia
Brief Title: New Topical Treatment for Continued Pain After Shingles
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Biomedical Development Corporation (Industry)
Collaborators: National Institute of Arthritis and Musculoskeletal and Skin Diseases (NIAMS) (NIH); The University of Texas Health Science Center, Houston (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Treatment
Other Study IDs: R43AR052998 (NIH); 1R43AR052998-01 (NIH); HSC-MS-06-0352
Record Dates: First submitted 2007-09-10; First posted 2007-12-04 (Estimated); Last update posted 2011-08-31 (Estimated); Status verified 2011-08

CONDITIONS: Postherpetic Neuralgia
Keywords: Post-herpetic Neuralgia; Pain after Shingles; Shingles; PHN
MeSH Terms: conditions — Neuralgia, Postherpetic; Herpes Zoster | interventions — Aspirin; Lidocaine; Anesthetics, Local

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- 1 (Experimental): Participants will receive one of three different topical treatments on Days 8, 15, or 22.
  Interventions: Drug: Epikeia coatings with aspirin; Drug: Epikeia coatings with lidocaine; Other: Epikeia coatings alone

INTERVENTIONS:
Drug: Epikeia coatings with aspirin — Applied to affected skin area using a roll-on ball applicator
  Other Names: Epikeia coatings with acetylsalicylic acid
Drug: Epikeia coatings with lidocaine — Applied to affected skin area using a roll-on ball applicator
  Other Names: Epikeia coatings with local anesthetic
Other: Epikeia coatings alone — Applied to affected skin area using a roll-on ball applicator

SUMMARY:
Shingles is an outbreak of rash or blisters on the skin that is caused by the same virus that causes chicken pox. Some people experience continued pain even after the shingles rash and blisters have healed; this pain is known as postherpetic neuralgia. The purpose of this study is to evaluate the effectiveness of a new topical treatment for postherpetic neuralgia in adults.

DETAILED DESCRIPTION:
After an initial infection of chicken pox, the varicella-zoster virus can remain dormant inside nerve cells. Years later, the virus can be reactivated, causing a repeat outbreak called shingles. The first symptom of shingles is usually a burning or tingling pain in one particular location and on one side of the body. This pain can range from mild to severe. Other possible symptoms of shingles include numbness and itching. After several days or 1 week, a rash of fluid-filled blisters similar to chicken pox appears. For most healthy people, a case of shingles heals within a month. However, some people continue to feel pain after the rash and blisters have resolved; this pain is known as postherpetic neuralgia. Current treatments for postherpetic neuralgia include antiviral drugs, steroids, antidepressants, anticonvulsants, and topical products. A new topical treatment consists of a liquid product that is applied directly to the skin to let dry and form a thin, transparent barrier film. In contrast to creams or ointments that can stay in contact with skin for only minutes, this product remains intact on the skin for many hours, providing sustained delivery of a drug or medication while maintaining barrier protection for the skin. The purpose of this study is to evaluate the effectiveness of this new topical treatment for postherpetic neuralgia in adults.

This study will last about 3 weeks and will include seven study visits on Days 1, 8, 9, 15, 16, 22, and 23. All study visits will include questionnaires on pain levels and an examination and digital photos of the affected skin area. The study visit on Day 1 will also include a urine pregnancy test and a review of medical and medication history. During the study visits on Days 8, 15, and 22, one of three topical products will be applied to participants' affected skin. The product will dry on the skin in 30 to 45 seconds. Participants will then wait at the study site for 1.5 hours, after which they will record the time when they experienced pain relief. At each of these three treatment visits, participants will receive one of the following three topical products: Epikeia coatings with aspirin, Epikeia coatings with local anesthetic, and Epikeia coatings alone. At these three study visits, questionnaires, examinations, and digital photographs will occur both before and after the products are applied to the skin. Throughout the study, participants will record their pain levels and medications in a diary, which will be reviewed at all study visits.

ELIGIBILITY:
Inclusion Criteria:

* In good general health
* Postherpetic neuralgia, defined as pain persisting more than 4 months after onset of herpes zoster outbreak
* Willing to use effective forms of contraception for the duration of the study

Exclusion Criteria:

* Known lidocaine sensitivity or allergy
* Inability to discontinue use of any nonstudy lidocaine-containing products for the duration of the study
* Known hypersensitivity to aspirin
* Open herpes zoster blisters
* Known sensitivity or allergy to an amide-type local anesthetic agent
* Existing conditions that make participation unsafe
* Pregnant
* Immunocompromised (e.g., HIV infected)
* Herpes zoster in any dermatome (area of skin innervated by a specific sensory nerve) affecting the face or scalp
* Affected skin area is greater than 420 square cm
* Affected area includes skin breakdown or nonintact skin
* Affected area consists of more than one contiguous area

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2006-09; Primary Completion 2008-08 (Actual); Study Completion 2008-09 (Actual)

PRIMARY OUTCOMES:
Latency to analgesia onset and duration of analgesia measures | Between 8 and 16 hours after treatment application

SECONDARY OUTCOMES:
Skin irritation potential | Between 8 and 24 hours after treatment application

CONTACTS AND LOCATIONS:
Overall Officials: Adelaide A. Hebert, MD, Principal Investigator — The University of Texas Health Science Center, Houston
Locations (1):
- Dermatology Clincial Reseach Center, Houston, Texas, United States